CLINICAL TRIAL: NCT07117994
Title: Radicle Revive™ 24_VPH: A Randomized, Double-Blind, Placebo-Controlled, Direct-to-Consumer Trial Assessing the Impact of Health and Wellness Products on Hormonal Health and Associated Health Outcomes in Women With Peri-Menopausal Health Issues
Brief Title: Radicle Revive 24: A Study of Health and Wellness Products on Hormonal Health and Associated Health Outcomes in Women With Peri-Menopausal Health Issues
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radicle Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RADX_P_2414_VPH
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-07

CONDITIONS: Stress; Menopause; Fatigue; Sleep
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Intervention Model Description: Participants will be stratified then randomized to one of the study arms. Each participant will have an equal chance of being assigned to each study arm.
Who Masked: Participant, Investigator
Masking Description: The investigator is blinded to the participants' assigned study products. Participants are blinded to the study product they received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Control 1 (Placebo Comparator): Radicle Revive Placebo Control Form 1
  Interventions: Dietary Supplement: Radicle Revive Placebo Control Form 1
- Active Product 1 (Experimental): Radicle Revive Active Study Product 1
  Interventions: Dietary Supplement: Radicle Revive Active Study Product 1

INTERVENTIONS:
Dietary Supplement: Radicle Revive Placebo Control Form 1 — Participants will use their Placebo Control Form 1 as directed for a period of 6 weeks.
  Arms: Placebo Control 1
Dietary Supplement: Radicle Revive Active Study Product 1 — Participants will use their Radicle Revive Active Study Product 1 as directed for a period of 6 weeks.
  Arms: Active Product 1

SUMMARY:
A Randomized, Double-Blind, Placebo-Controlled, Direct-to-Consumer Trial Assessing the Impact of Health and Wellness Products on Hormonal Health and Associated Health Outcomes in Women with Peri-Menopausal Health Issues

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study conducted with adult participants, residing in the United States.

Eligible participants (1) are females, (2) have peri-menopausal-related health issues for 3 months or longer, (3) have the opportunity to improve by at least 30% in the primary outcome, and (4) express acceptance in taking study products and not knowing the formulation identities until the end of the study.

Participants that report a known cardiac dysfunction, liver or kidney disease may be excluded. Participants that report a known contraindication or with well-established, significant safety concerns due to illness will be excluded. Heavy drinkers and ag who are pregnant or breastfeeding will be excluded. Participants that report taking medications with a known contraindication or with well-established, significant safety concerns will be excluded.

Self-reported data are collected electronically from eligible participants for 7 weeks. Participant reports of health indicators will be collected at baseline, throughout the active period of study product use, and in a final survey. All study assessments will be electronic; there are no in-person visits or assessments for this real-world evidence study.

ELIGIBILITY:
Inclusion Criteria:

* Adults, at least 40 years of age at the time of electronic consent, inclusive of all ethnicities, races, and gender identities
* Assigned sex at birth is female
* Resides in the United States
* Identifies menstrual status as perimenopausal
* Has the opportunity for at least 30% improvement in their primary health outcome
* Indicates having peri-menopausal issues for 3 months or longer
* Expresses a willingness to take a study product and not know the product identity (active or placebo) until the end of the study

Exclusion Criteria:

* Individuals who report any of the following during screening will be excluded from participation:
* Reports being pregnant or breastfeeding
* Unable to provide a valid US shipping address and mobile phone number
* Reports current enrollment in another clinical trial
* Reports being a heavy drinker (defined as drinking 3 or more alcoholic beverages per day)
* Unable to read and understand English
* Reports a current and/or recent (up to 3 months ago) major illness and/or surgery that poses a known, significant safety risk.
* Reports a diagnosis of cardiac dysfunction, liver or kidney disease that presents a known contraindication and/or a significant safety risk with any of the study product ingredients.
* NYHA Class III or IV congestive heart failure, atrial fibrillation, uncontrolled arrhythmias, cirrhosis, end-stage liver disease, stage 3b or 4 chronic kidney disease, or kidney failure
* Reports taking medications that have a well-established moderate or severe interaction, posing a substantial safety risk with any of the study product ingredients.
* Anticoagulants, antihypertensives, anxiolytics, antidepressants, chemotherapy, immunotherapy, sedative hypnotics, medications that warn against grapefruit consumption, corticosteroids at doses greater than 5 mg per day, diabetic medications, oral anti-infectives (antibiotics, antifungals, antivirals) to treat an acute infection, antipsychotics, MAOIs, or thyroid products
* Reports current use of the primary ingredient(s) and/or similar product(s) to the active study product(s) that may limit the effects of the study products and/or pose a safety risk to participants
* Reports an allergy to and/or disinterest in any of the possible study product ingredients
* Lack of reliable daily access to the internet

Ages: 40 Years to 105 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2025-08-05 (Actual); Primary Completion 2025-11-12 (Actual); Study Completion 2025-11-12 (Actual)

PRIMARY OUTCOMES:
Change in Perceived Stress | 6 weeks
  Change in perceived stress: Difference between rates of change over time in Perceived Stress score as assessed by NIH Toolbox Perceived Stress Survey (scale 10-50; where the higher scores correspond to worse perceived stress)

SECONDARY OUTCOMES:
Change in General Menopausal Health | 6 weeks
  Change in other menopausal health issues: Other menopausal health issues assessed by Radicle General Menopausal Health Issues (Point range: 6 - 68; where higher scores correspond to more severe menopausal health issues)
Change in Sleep Disturbance | 6 weeks
  Change in sleep: Difference in rates of change over time in sleep score as assessed by PROMIS Sleep Disturbance 8A (scale 8-40; where higher scores correspond to higher levels of sleep disturbance)
Change in Fatigue | 6 weeks
  Change in fatigue: Difference in rates of change over time in fatigue score as assessed by Patient Reported Outcome Measurement System (PROMIS) Fatigue 8A (scale 8-40; where higher scores correspond to more severe fatigue)
Minimal clinically important difference (MCID) in perceived stress | 7 weeks
  Likelihood of experiencing minimal clinically important difference in perceived stress, as assessed by NIH Toolbox Perceived Stress Survey (scale 10-50; where the higher scores correspond to worse perceived stress)
Minimal clinically important difference (MCID) in menopausal health issues | 7 weeks
  Likelihood of experiencing minimal clinically important difference in menopausal health issues score assessed by Radicle General Menopausal Health Issues (Point range: 6 - 68; where higher scores correspond to more severe menopausal health issues)
Minimal clinically important difference (MCID) in fatigue | 7 weeks
  Likelihood of experiencing minimal clinically important difference in fatigue score as assessed by PROMIS Fatigue 8A (scale 8-40; where higher scores correspond to more severe fatigue)
Minimal clinically important difference (MCID) in sleep | 7 weeks
  Likelihood of experiencing minimal clinically important difference in sleep score as assessed by PROMIS Sleep Disturbance 8A (scale 8-40; where higher scores correspond to higher levels of sleep disturbance)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Hewlings, Principal Investigator — Radicle Science Inc.
Locations (1):
- Radicle Science, Inc, Del Mar, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with researchers outside of Radicle Collaborators on this study.

REFERENCES:
- See also: Related Info — https://www.radiclescience.com